CLINICAL TRIAL: NCT03011853
Title: Survival After Failure of First-line Non-invasive Ventilation in Acute on Chronic Obstructive Pulmonary Disease: a Cohort Study of Intensive Care Patients.
Brief Title: Survival After Failed First-line Non-invasive Ventilation in Acute on Chronic Obstructive Pulmonary Disease
Status: Completed | Type: Observational
Sponsor: Swedish Intensive Care Registry (Other)
Responsible Party: Sponsor
Other Study IDs: NIV4COPD
Record Dates: First submitted 2016-11-20; First posted 2017-01-05 (Estimated); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Chronic Obstructive Airways Disease Exacerbated; Critical Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Non-invasive only: Non-invasive ventilation as first and only respiratory support
  Interventions: Procedure: Non-invasive and/or invasive mechanical ventilation
- Invasive: Invasive ventilation with intubation as first respiratory support
  Interventions: Procedure: Non-invasive and/or invasive mechanical ventilation
- NIV+Inv: Non-invasive ventilation as first respiratory support followed by invasive ventilation with intubation
  Interventions: Procedure: Non-invasive and/or invasive mechanical ventilation

INTERVENTIONS:
Procedure: Non-invasive and/or invasive mechanical ventilation — Use of Non-invasive and invasive mechanical ventilation, focussing particularly on the first respiratory support mode in ICU

SUMMARY:
Observational cohort study of mid-to-long term survival of patients with acute on chronic obstructive pulmonary disease, analyzed per type of ventilation support provided during first 24 hours in intensive care.

DETAILED DESCRIPTION:
Registry setting and procedures:

The Swedish Intensive Care Registry (SIR) collects a comprehensive dataset of patient characteristics, intensive care procedures and outcomes using detailed guidelines.

Continuous data are collected as raw data, validated locally and transferred electronically to the registry for central validation (confirmed to be within prespecified limits and inconsistencies and illogical entries identified). If necessary, data are returned for correction and revalidation before being accepted and added to the master database.

Study participants:

Patients with COPD as the principal diagnosis during their ICU stay were included in the study cohort. When patients had multiple admissions during the study period due to COPD the last admission only was included. Patients were excluded when nursing workload scores indicated active ventilation support during the first 24 hours but information on type of support (non-invasive or invasive ventilation) was lacking. Participants with missing vital status were also excluded from analysis.

Patients were grouped according to the mode of the first-line ventilation support that was given during the initial 24 hours in ICU. The Standard therapy group did not receive any active ventilation support, the NIV only group received non-invasive ventilation support only, the NIV + Invasive mechanical ventilation (IMV) group received NIV followed by intubation and invasive ventilation support and, the IMV group were intubated and received invasive ventilation support without any preceding NIV trial.

ELIGIBILITY:
Inclusion Criteria:

* Principal diagnosis of ICU stay: Acute on Chronic Obstructive Pulmonary Disease

Exclusion Criteria:

* Multiple admissions of patients during study period: every admission but the last one is excluded.
* Conflicting data on ventilation support
* Vital status missing at 6 months

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients admitted to ICUs that are members of the Swedish Intensive Care Registry and participate in data collection and audit.
Sampling Method: Non-Probability Sample
Enrollment: 7900 (Actual)
Dates: Start 2008-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Six month survival | 180 days
  180 days beginning with the day of admission to ICU

SECONDARY OUTCOMES:
One year survival | 365 days
  365 days beginning with the day of admission to ICU
ICU length of stay | up to 180 days
  From time of admission to time of discharge or death, assessed up to 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Sten M Walther, MD PhD, Principal Investigator — Linkoeping University
Locations (1):
- Västerviks sjukhus, Västervik, Sweden

IPD SHARING:
Plan to Share IPD: No